CLINICAL TRIAL: NCT06115161
Title: Development and Validation of an Instrumented Ankle-foot Orthosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The instrumented orthosis prototype was never finished.
Sponsor: TOPMED (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Turbomed Orthotics Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 241_Tur_ApEval
Record Dates: First submitted 2023-09-13; First posted 2023-11-02 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Foot Drop
Keywords: ankle foot orthosis; validation; survey; gait analysis; biomecanics
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Intervention Model Description: Trial with condition crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait Analysis (Experimental): Gait analysis with the instrumented orthosis as well as a reference sysmtem (Vicon Vantage 5).
  Interventions: Device: Instrumented Orthosis

INTERVENTIONS:
Device: Instrumented Orthosis — Gait analysis will be performed with the instrumented orthosis as well as the reference system.

SUMMARY:
Foot drop (weakness or paralysis of the muscles that lift the foot) refers to a condition that prevents people from properly lifting their foot and toes while walking. Foot drop has a negative impact on the balance, mobility, and confidence of people with the condition. Dragging one's toes on an uneven floor or a carpet can lead to tripping and falling.

TurboMed Orthotics Inc. has developed various orthoses for several years in order to improve the gait and quality of life for people suffering from foot drop. In order to help clinicians better monitor and assess gait parameters over time, the company wants to offer clinicians a tool for a more rigorous analysis. Thus, the objective of the proposed project is to develop a questionnaire for identifying the clinical need for the data generated by the instrumented orthosis. The instrumented orthosis will also be compared to a reference system in a validation effort.

ELIGIBILITY:
Inclusion Criteria for Patients questionnaire:

* Having foot drop

Inclusion Criteria for Clinician questionnaire:

* Being a clinician who treats foot drop patients

Inclusion Criteria for Gait analysis:

* Having foot drop

Exclusion Criteria for Gait analysis:

* Not being able to walk without a cane or a walker
* Having lower extremity spasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Gait Temporal parameters | During the intervention, 10 walking trials will be assessed, all trials will be performed in the same session
  Gait Temporal parameters measured by the instrumented orthosis and the reference system, in seconds, these include the different phase durations(stride, stance and swing).
Heel strike angle | During the intervention, 10 walking trials will be assessed, all trials will be performed in the same session
  Heel strike angle measured by the instrumented orthosis and the reference system
Gait Spatial parameters | During the intervention, 10 walking trials will be assessed, all trials will be performed in the same session
  Gait Spatial parameters measured by the instrumented orthosis and the reference system, in meters, these include the length and width of the stride.
Gait speed | During the intervention, 10 walking trials will be assessed, all trials will be performed in the same session
  Gait speed measured by the instrumented orthosis and the reference system, in meters per second.

CONTACTS AND LOCATIONS:
Locations (1):
- TOPMED, Québec, Canada

IPD SHARING:
Plan to Share IPD: No